CLINICAL TRIAL: NCT03787069
Title: Effect of Intravenous Lignocaine vs Placebo on Hemodynamic Response During Intubation
Brief Title: Intravenous Lignocaine vs Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indus Hospital and Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRD_IRB_2017_07_002
Record Dates: First submitted 2018-12-24; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Hemodynamic Stability Post Intubation in Laryngoscopy Surgery

STUDY DESIGN:
Intervention Model Description: Equal allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lignocaine group (Experimental): This group will be given 1.5 mg/kg I/V lignocaine before intubation
  Interventions: Drug: iv Lignocaine vs placebo
- Placebo (Placebo Comparator): This group will be given 6 ml normal saline before intubation
  Interventions: Drug: iv Lignocaine vs placebo

INTERVENTIONS:
Drug: iv Lignocaine vs placebo — Lignocaine is available in an ampule of 10 ml containing 20 mg/ml of lignocaine or 2%, Lignocaine will be given in dose of 1.5 mg/kg I/V

SUMMARY:
To assess the mean hemodynamic responses post-intubation in patients given intravenous lignocaine pre-intubation as compared to a placebo pre-intubation in patients undergoing laryngoscopy surgery

DETAILED DESCRIPTION:
After identifying the candidate, details will be carefully discussed with the subject. The subject (or, when necessary, the parent or legal guardian if the subject is younger than 18 years of age or under guardianship) will be read the approved protocol consent form. Patients who have given informed consent to participate in the study will be randomized into one of the two study arms one day before the procedure. The study team present will open the sealed envelopes provided by the Indus Hospital Research Center's Clinical Research Unit (CRU) that provides the study arm allocation. The envelopes will follow the SNOSE protocol.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II
* Age 20-60 years
* Mallampatti , II
* All surgeries are done under GA
* Both genders
* Those patients giving informed consent

Exclusion Criteria:

* Difficult airway assessed during pre-op anaesthesia assessment
* Unanticipated difficult airway based on the previous history of difficult intubation
* BMI >30,
* Micrognathia and microglossia based on pre-op anaesthesia assessment,
* Diabetic patient with autonomic dysfunction liver disease, cardiovascular disease, pheochromocytoma, Cushing syndrome
* Patients who do not give informed consent

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
MAP | post-intubation 3 minutes to 10 minutes
  mean arterial pressure
Pulse | post-intubation 3 minutes to 10 minutes
  Heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- The Indus Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided